CLINICAL TRIAL: NCT04668807
Title: Assessment of the Technical Capabilities of the "SMART ANGEL" Intra-hospital System 's Connected Medical Device (CMD)
Brief Title: Technical Capabilities of the "SMART ANGEL Intra-hospital" System 's Connected Medical Device (CMD)
Acronym: SMART-METRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Evolucare Technologies (Industry); InES - Innovation Electronic Software (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: APHP190708; 2019-A02197-50 (Other: N° IDRCB)
Record Dates: First submitted 2020-11-05; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-02

CONDITIONS: Medical Device
Keywords: Connected Medical Device; Device Feasibility; Post-operative mortality; "SMART ANGEL intra-hospital" system

STUDY DESIGN:
Intervention Model Description: Measurement of 3 constants (SpO2, heart rate and respiratory rate) in patients with a non-ambulatory surgical or interventional act lasting more than 2 hours whose constants are monitored by the reference device in the operating room and the Connected Medical Device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected Medical Device (Experimental): "SMART ANGEL Intra-hospital" System 's Connected Medical Device (DMC) measuring physiological parameters in the operating room
  Interventions: Device: Connected Medical Device
- Traditional system (Active Comparator): Traditional wired transmission system between the sensor and the data processing device in the operating room
  Interventions: Device: Traditional transmission system

INTERVENTIONS:
Device: Connected Medical Device — Monitoring of three simple physiological parameters (SpO2, heart rate and respiratory rate) with a Connected Medical Device (DMC) in the operating room
  Arms: Connected Medical Device
Device: Traditional transmission system — Monitoring of physiological parameters with a traditional wired transmission system between the sensor and the data processing device in the operating room
  Arms: Traditional system

SUMMARY:
Post-operative mortality in case of scheduled surgery is 3% in France (Lancet 2013) mainly due to cardiovascular or respiratory complications, by decompensation of pre-existing pathologies.

Complications due to the medical practice are the third cause of morbidity(BMJ, 2016). More than half are preventable and are mainly observed in surgical patients. In conventional hospitalization, excluding intensive care, monitoring is done discontinuously for most of the patients, which does not allow early diagnosis of a vital cardiovascular or respiratory failure.

Diagnosis and late treatment do not allow good recovery. The early identification of a vital failure by the continuous monitoring of three simple physiological parameters (SpO2, heart rate and respiratory rate) would allow faster management by the hospital staff and a reduction in immediate and possibly delayed postoperative mortality.

DETAILED DESCRIPTION:
The challenge of this research is to transpose in an ordinary hospitalization unit the continuous monitoring of vital functions carried out in intensive care by the continuous measurement of simple parameters using a Connected Medical Device (CMD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients receiving a non-ambulatory surgical or interventional procedure lasting more than 2 hours
* Affiliation with a social security syste, beneficiarie or eligible people (excluding State Medical Assistance (AME))
* Written consent of the patient

Exclusion Criteria:

* Patient carrying a multi-resistant germ and placed in isolation
* Patient's known linguistic inability to understand the study
* Non-ambulatory surgical or interventional act in an emergency situation
* Patients under legal protection : curatorship or guardianship
* Known pregnancy or nursing woman
* Patients with implantable cardiac pacemakers, implantable defibrillators or neurostimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Agreement between the values measurements produced by the traditional monitoring system in the operating theater and the connected medical device of the "SMART ANGEL intra-hospital" system | at 2 hours

SECONDARY OUTCOMES:
Evaluation of missing data due to device malfunction | at 2 hours
Nurse satisfaction (System Usability Scale) | at 2 hours
Occurrence of events during the course of the study | at 2 hours
Time needed by the nursing staff to set up the system | at 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MARTY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France